CLINICAL TRIAL: NCT01611987
Title: The Role of Exercise in Modifying Outcomes for People With Multiple Sclerosis
Acronym: MStep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Mayo, PhD, Principal Investigator, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR258309; NCT01032707 (obsolete NCT alias)
Record Dates: First submitted 2012-05-22; First posted 2012-06-05 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSTEP (Experimental): The MSTEP program is a 6 day tailored exercise program. It includes flexibility, aerobic, peripheral strengthening, core and balance training, power and speed training and push days.
  Interventions: Other: MStep
- General guideline approach (Active Comparator): The general Guideline approach is the general guidelines that are recommended for people with MS by the Canadian Society Exercise Physiology.
  Interventions: Other: General guideline approach

INTERVENTIONS:
Other: MStep — Participant will meet with instructor twice to learn how to exercise safely. Exercises will be demonstrated and practiced under the direct supervision of the instructor. Written details and pictures will be made. Variety in exercise will be encouraged to promote long-term adherence. Stretching, strengthening and relaxation exercises will be given. Persons will be given Thera Band® to facilitate resistance exercise training and instructed how to progress. Equipment such as Nordic Walking Poles, stationary bicycle, BOSU®, or exercise balls will be available. Rather than having a fixed rigid prescription, the aim is to get people to intuitively adjust the amount of resistance so they feel they are working without causing harm, they are not doing the same boring activity, week in week out.
  Arms: MSTEP
Other: General guideline approach — Individuals in the control condition will meet with the exercise instructor on two occasions during the first two weeks to review key components of public health guidelines for physical activity and health. In brief, the general guidelines for MS are (i) aerobic and endurance exercise for 30 minutes per session, 3 times per week at an intensity of 60% to 75% of heart rate peak; (ii) weight training for weak muscles, 2 days per week, on non-endurance days, 8 to 15 repetitions per exercise; and (iii) stretching daily with active or passive range of motion exercises, or attendance at Yoga or Tai Chi classes.
  Arms: General guideline approach

SUMMARY:
Despite the benefits of exercise and physical activity people with Multiple Sclerosis (MS) are relatively inactive. Physical activity is important for persons with disabilities to maintain physical function. A lack of physical activity can contribute to heart disease, osteoporosis, obesity, and diabetes. At the moment, the best way for people with MS to exercise and be physical activity is unknown. People with MS report not knowing what to do. This is a barrier to exercise.

The global aim of this study is to contribute evidence for the role of targeted exercise in altering MS outcomes over time. The design is a randomized controlled trial (RCT). The primary research question is to what extent does an MS Tailored Exercise Program (MSTEP) result in greater improvements in exercise capacity and related outcomes in comparison to a program based on general guidelines for exercise among people with MS who are sedentary and wish to engage in exercise as part of MS self-management. The primary outcome for this question is exercise capacity measured using cycle ergometry. However exercise efficiency, functional ambulation, strength, components of quality of life including frequency and intensity of fatigue symptoms, mood, global physical function, health perception, and illness intrusiveness, will also be measured as components of a global response outcome. The first confirmatory hypothesis is that MSTEP will result in a greater proportion of people making clinically relevant gains (at least 10% change) in exercise capacity than with general guidelines after 12 months of intervention; a secondary hypothesis is that, while there may be some decline in exercise capacity among individuals from end of intervention to follow-up one year later, the decline will be greater in the general guideline group augmenting the difference between groups in the proportion making 10% change from study entry to 24 months. In other words, gains will be maintained more for the MSTEP group over the general guideline group.

An exploratory hypothesis is that more of the targeted outcomes will improve with the MSTEP program than the general guideline approach. An explanatory hypothesis is that these gains will be accompanied by reports of greater exercise enjoyment and exercise self-efficacy (confidence) with the MSTEP program than with the general guideline program leading to more consistent exercise engagement and improved long-term adherence.

DETAILED DESCRIPTION:
The proposal is for an assessor-blind, parallel-group, stratified, randomized controlled trial. Potential participants will be identified from the population of persons enrolled in 3 MS clinics in the Montreal area and in 3 clinics in Toronto. All persons who are known to be ambulatory and not to have co-morbidity preventing exercise engagement or capacity to consent will be informed of the study in writing and will be invited for an assessment to determine eligibility for entry into the trial. Those consenting will be randomly assigned to either the MSTEP program or the general exercise guideline program. The intervention period will be one year with follow-up to a second year.

The investigators are targeting a sample size of 120 per group (total 240), which would be sufficient to detect RR of > 1.5 with 80% power. Sample size estimated using pc-size software. The sample size takes into account that drop-outs will inflate the variance of outcomes as multiple imputation will be used to deal with missing data.

The main analysis will be logistic regression to test the main hypothesis related to the superiority of the MSTEP program based on a greater proportion of people making a clinically relevant gain in exercise capacity at 1 year. A secondary outcome will be the differences in proportions at 2 years also using logistic regression. The analysis will be based on intention-to-treat and all persons will be analysed in the groups to which they were randomized.

A secondary analysis will estimate the impact of exercise on the other relevant outcomes. For this approach, each outcome will be converted to a binary response variable based on published clinically meaningful changes and generalized estimating equations (GEE) will be used to test the rate of response in the MSTEP program to the rate of response in the general guideline approach. Multiple outcomes improves the efficiency of the study as the total number of data points is equivalent to the total n multiplied by the number of tests and reduced by the extent to which the outcomes are correlated. Highly correlated outcomes will make the effective sample size smaller than less strongly correlated outcomes. If there is a statistically significant effect of the intervention, then and only then, can the effects of the separate outcomes be interpreted as real.

The results of the trial will be used to develop guidelines for exercise for MS. The investigators are in the process of copyrighting the name of the program (MSTEP). Upon publication of the findings, the description of content will be made available at no cost. If proven effective, a training guide for professionals and patients will be produced most likely taking advantage of the end-of-grant Knowledge Translation (KT) Supplement. Note: The investigators have been funded by the KT supplement to produce a general guide for people with MS, entitled: Getting on with Your Life with MS. The knowledge generated can be used by people with MS and health professional to promote exercise engagement.

ELIGIBILITY:
Inclusion Criteria:

* be community dwelling individuals aged 19 -65 who have been diagnosed after 1994 with MS or CIS;
* be able to speak and read English or French;
* be capable of walking 100 meters without a walking aid (EDSS ≤ 5.5), even if they do use an aid for daily activities.

Exclusion Criteria:

* have an additional illness that restricts their function; and/or
* had suffered at least one relapse during the past 30 days (as defined by Polman) as this may affect physical activity/exercise participation.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
oxygen consumption | 3 timepoints: baseline, at 12 monts, at 24 months
  VO2peak will be determined using an incremental graded cycle ergometer test. Greater oxygen consumption implies in better exercise capacity

SECONDARY OUTCOMES:
muscle strength measured with Biodex | 3 timepoints: Baseline, at 12 months, at 24 months
  Greater values imply greater muscle strength
6 Minute Walk test (6MWT) | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  Distance walked will be measured with the 6-Minute Walk Test. Greater values imply that a longer distance was covered within 6 minutes
Anaerobic leg power | 1 timepoint: baseline
  Greater value indicate greater anaerobic leg power
Patient Determined Disease Steps (PDDS) | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  Patient Determined Disease Steps (PDDS) is a scale focusing mainly on how well someone walk. It ranges from mild symptoms that do not affect physical activity to inability to sit in a wheel chair for more than 1 hour.
Change in fatigue levels | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  Fatigue will be measured with a single item question asking them the number of days that they felt certain levels of fatigue.
Rand 36 | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  Health status will be measured with the Rand36 Health Status Survey. The Rand36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.
EQ-5D | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  The respondent is asked to indicate his/her health state in each of 5 dimensions. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents
Patient generated Index | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  Participants will be asked to identify 5 most important areas of their life that are affected by multiple sclerosis. A second step will be to score how much affected these identified areas were over the past MONTH, in a scale from 1 to 10.
Exercise Self-Efficacy Scale | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  This will be measured by the Exercise Self-Efficacy Scale, in which participants are asked how certain they are that they can get to perform an exercise routine regularly (three or more times a week). The scale ranges from 0 (not confident) to 100 (highly confident).
Change in perception about exercise benefits and exercise barrier | 5 timepoints: at baseline, at 6 months, at 12 months, at 18 months, at 24 months
  It will be measured with a self-reported questionnaire. For the exercise benefits, the scale range as "strongly disagree, disagree, agree, strongly agree".
  For the exercise barriers the scale range as "sometimes a barrier", "often a barrier"
Modified Canadian Aerobic Fitness test | 3 timepoints: 3 month, 6 month and 18 month
  mCAFT is a graded step test and can predict VO2peak using a regression equation recently published. Thus, we are confident that we will get usable data for each person and as we are looking for a proportion of people who change over time, persons who do not achieve a peak and have low values on the mCAFT will have a very low value for exercise capacity.
  Greater steps cadence imply on greater oxygen cost

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Mayo, PhD, Principal Investigator — McGill University
Locations (5):
- Canada (5):
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Rehabiliation Institute, Toronto, Ontario
  - CHUM, Montreal, Quebec
  - Muhc - Mnh, Montreal, Quebec

REFERENCES:
- [Background] Warren S, Warren KG. Prevalence, incidence, and characteristics of multiple sclerosis in Westlock County, Alberta, Canada. Neurology. 1993 Sep;43(9):1760-3. doi: 10.1212/wnl.43.9.1760. PMID 8414027
- [Background] Warren S, Warren KG, Svenson LW, Schopflocher DP, Jones A. Geographic and temporal distribution of mortality rates for multiple sclerosis in Canada, 1965-1994. Neuroepidemiology. 2003 Jan-Feb;22(1):75-81. doi: 10.1159/000067111. PMID 12566957
- [Background] Turner AP, Kivlahan DR, Haselkorn JK. Exercise and quality of life among people with multiple sclerosis: looking beyond physical functioning to mental health and participation in life. Arch Phys Med Rehabil. 2009 Mar;90(3):420-8. doi: 10.1016/j.apmr.2008.09.558. PMID 19254606
- [Background] Poppe AY, Wolfson C, Zhu B. Prevalence of multiple sclerosis in Canada: a systematic review. Can J Neurol Sci. 2008 Nov;35(5):593-601. doi: 10.1017/s0317167100009380. PMID 19235443
- [Background] White LJ, Castellano V. Exercise and brain health--implications for multiple sclerosis: Part 1--neuronal growth factors. Sports Med. 2008;38(2):91-100. doi: 10.2165/00007256-200838020-00001. PMID 18201113
- [Background] White LJ, Castellano V. Exercise and brain health--implications for multiple sclerosis: Part II--immune factors and stress hormones. Sports Med. 2008;38(3):179-86. doi: 10.2165/00007256-200838030-00001. PMID 18278981
- [Background] Dalgas U, Stenager E, Ingemann-Hansen T. Multiple sclerosis and physical exercise: recommendations for the application of resistance-, endurance- and combined training. Mult Scler. 2008 Jan;14(1):35-53. doi: 10.1177/1352458507079445. Epub 2007 Sep 19. PMID 17881393
- [Background] Mayo N. Setting the agenda for multiple sclerosis rehabilitation research. Mult Scler. 2008 Nov;14(9):1154-6. doi: 10.1177/1352458508096567. No abstract available. PMID 18952830
- [Background] Motl RW, Snook EM, McAuley E, Gliottoni RC. Symptoms, self-efficacy, and physical activity among individuals with multiple sclerosis. Res Nurs Health. 2006 Dec;29(6):597-606. doi: 10.1002/nur.20161. PMID 17131278
- [Background] Motl RW, McAuley E, Snook EM. Physical activity and multiple sclerosis: a meta-analysis. Mult Scler. 2005 Aug;11(4):459-63. doi: 10.1191/1352458505ms1188oa. PMID 16042230
- [Background] Rietberg MB, Brooks D, Uitdehaag BM, Kwakkel G. Exercise therapy for multiple sclerosis. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003980. doi: 10.1002/14651858.CD003980.pub2. PMID 15674920
- [Background] Asano M, Dawes DJ, Arafah A, Moriello C, Mayo NE. What does a structured review of the effectiveness of exercise interventions for persons with multiple sclerosis tell us about the challenges of designing trials? Mult Scler. 2009 Apr;15(4):412-21. doi: 10.1177/1352458508101877. PMID 19324979
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Hayes HA, Gappmaier E, LaStayo PC. Effects of high-intensity resistance training on strength, mobility, balance, and fatigue in individuals with multiple sclerosis: a randomized controlled trial. J Neurol Phys Ther. 2011 Mar;35(1):2-10. doi: 10.1097/NPT.0b013e31820b5a9d. PMID 21475078
- [Derived] Mayo NE, Bayley M, Duquette P, Lapierre Y, Anderson R, Bartlett S. The role of exercise in modifying outcomes for people with multiple sclerosis: a randomized trial. BMC Neurol. 2013 Jun 28;13:69. doi: 10.1186/1471-2377-13-69. PMID 23809312
- See also: Multiple Sclerosis Society of Canada — http://www.mssociety.ca.